CLINICAL TRIAL: NCT06495268
Title: Healthy Hearing for Healthy Ageing: a Proof-of-concept Randomized Controlled Trial of Data-driven Hearing Rehabilitation Versus Standard Care in Older Adults with Hearing Impairment.
Brief Title: Healthy HeaAring for Healthy Ageing: Data-driven Hearing Rehabilitation Intervention to Promote Healthy Hearing
Acronym: HAHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KUH5551893
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Sensorineural Hearing Loss; Cognitive Decline
Keywords: Hearing Impairment; Hearing Rehabilitation; Hearing Loss; Cognition; Data-driven rehabilitation
MeSH Terms: conditions — Hearing Loss, Sensorineural; Cognitive Dysfunction; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either intervention (individualised data-driven hearing rehabilitation) or control group (standard care hearing rehabilitation) by computer-generated allocation in blocks of four (two individuals randomly allocated to each group).
  The intervention group will receive individually fitted HAs with immediate SPIN-based benefit validation. HA selection and individual tailoring will also be based on hearing questionnaires data. Participants are invited to intervention-related monitoring appointments at 3, 6 and 12 months.
  The control group will receive the same HAs fitted according to the standard care protocol. Standard care follow-up includes a phone call check 3 months after the primary fitting. Additional monitoring/re-fitting may be offered based on the participant's feedback and hearing rehabilitator's clinical judgement.
  12-month and 24-months follow-up appointments are arranged for both groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: By default, hearing rehabilitators will be aware of which group of participants they are assigned to, since those assigned to the intervention group will need to implement a HA fitting protocol different from standard care. Participants will not be actively told which group they are assigned to following randomisation, although complete masking may not be feasible based on the differences between HA fitting protocols. Outcome assessors, the PI, co-PI, and other key project team members will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualised data-driven hearing rehabilitation (Active Comparator): Participants in the intervention group will receive data-driven, regularly controlled hearing aid rehabilitation that is not part of the standard care protocol.
  Interventions: Other: Individualised data-driven hearing rehabilitation
- Standard care hearing rehabilitation (Active Comparator): The participants in the control group will receive the standard care HA rehabilitation currently conducted at the KUH Hearing Center.
  Interventions: Other: Standard care hearing rehabilitation

INTERVENTIONS:
Other: Individualised data-driven hearing rehabilitation — HA fittings will be conducted with the Real-Ear Measurements (REM) method that is recommended by the latest ISO-standard (21388:2020) and by the preliminary results of the BREM study at KUH. After the fitting of the HAs, participants' auditory-related outcomes will be immediately assessed using DigiKuulo and re-fitting is performed if needed based on the following criteria:
  1. The absolute improvement in the DIN test is less than 1,5dB (SNR), OR
  2. The absolute result of the DIN test is more than -8,5 dB (SNR) OR
  3. The participant is unsatisfied with the HA fitting
  Participants are invited to intervention-related monitoring appointments at 3, 6 and 12 months after the primary HA fitting. At these visits, auditory outcomes of the rehabilitation are assessed via DigiKuulo and re-fittings are performed as needed.
  Arms: Individualised data-driven hearing rehabilitation
Other: Standard care hearing rehabilitation — HA will be fitted with automatic algorithms by HA manufacturers and REM-fitting is only applied in complex cases based on the hearing rehabilitator's clinical judgement. Three months after the HA fitting, participants will be contacted via phone call to inquire about the status of the rehabilitation. Additional monitoring visits may be offered based on the participant's feedback. After the 3-month monitoring phone call participants will be advised to further contact the study team if they are dissatisfied with the amplification or for any other problem with their device.
  Arms: Standard care hearing rehabilitation

SUMMARY:
The goal of the HAHA trial is to prove that the treatment of HI and prevention of HI-related cognitive decline are most likely to be effective if HI is approached as a broader neurodegenerative entity with multifaceted manifestations currently unaddressed in clinical practice and managed using a novel individualised data-driven protocol for early hearing rehabilitation. The main hypothesis is that, compared with standard care, the data-driven rehabilitation will likely have broader benefits manifested in three key areas: hearing, cognition, and quality of life and psychosocial outcomes.

Participants will be randomized 1:1 to either intervention (individualised data-driven hearing rehabilitation) or control group (standard care hearing rehabilitation). The primary objective of this study is to investigate the effect of an optimized data-driven hearing rehabilitation protocol versus standard care protocol on change in speech perception in noise (SPIN) in older adults with mild to moderately severe sensorineural HI and without dementia.

DETAILED DESCRIPTION:
Hearing impairment (HI) is a major public health problem. HI has also been identified as a significant potentially modifiable risk factor for dementia. Thus, hearing rehabilitation may contribute to dementia risk reduction, although a causal HI-dementia relation is not fully established.

The HAHA trial will test an individualised, data-driven hearing rehabilitation protocol based on the ongoing BREM (Benefits of Real-Ear Measurement) study at KUH (clinicaltrials.gov ID NCT05621798). HAHA will use a pragmatic approach incorporated into routine specialized care (Hearing Center at the Dept of Otorhinolaryngology of KUH), to facilitate optimisation of the current HI clinical pathway and treatment process. This study is a proof-of-concept, single-site, 2-arm parallel group 12-month randomized controlled trial with a 12-month extended follow-up.

The investigators will recruite 200 participants referred to the Kuopio University Hospital Hearing Center from primary care that are aged 65 to 84 years with mild to moderately severe sensorineural HI and are about to receive their first HAs.

The intervention group will receive individually fitted HAs based on preliminary results from the ongoing BREM study at KUH to ensure adequate amplification, with immediate SPIN-based benefit validation. HA selection and individual tailoring will also be based on hearing questionnaires data. Participants are invited to intervention-related monitoring appointments at 3, 6 and 12 months after the primary HA fitting.

The control group will receive the same HAs fitted according to the standard care protocol. Standard care follow-up includes a phone call check 3 months after the primary fitting. Additional monitoring/re-fitting may be offered based on the participant's feedback and hearing rehabilitator's clinical judgement.

A range of auditory, cognitive, quality of life and psychosocial measures as well as exploratory measures such as EEG, MRI and vision-related measures are assessed at 12-month and 24-month visits on both groups. These assessments are included to investigate potential mechanisms underlying associations between HI, hearing rehabilitation, vision and cognition. The overall duration of the this trial is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderately severe sensorineural HI (PTA (0,5-4kHz) between 20-64 dB (HL), as per Global Burden of Disease Expert Group on Hearing loss criteria)
* Community-dwelling, i.e. living at home / not living in a care home or nursing home
* Proficiency in Finnish language
* First-time hearing aid user

Exclusion Criteria:

* Conductive hearing loss (air-bone gap more than 20 dB HL in two consecutive frequencies)
* Difference between hearing levels of the ears is more than 15dB (HL) in three consecutive frequencies
* Hearing aid contraindication
* Previously diagnosed dementia, or current use of cholinesterase inhibitors and/or memantine. If there is a current ongoing diagnostic process for suspected dementia, the decision on eligibility will be made by an experienced study physician based on medical records and clinical judgement.
* Any health conditions severely impairing vision, mobility, communication, and/or ability to participate in study visits and complete study assessments, as judged by the study nurse and/or physician.

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Finnish Matrix Sentence Test (FMST) | Change measures: 0 months, 12 months, 24 months
  A Speech-in-Noise test, validated for the Finnish language. In the test participants will listen to five-word sentences chosen out of a standardized and optimized word matrix under stationary background noise (65dB SPL). The result of the FMST is the signal-to-noise ratio (SNR) at which the participant identifies 50% of the presented word items correctly, this is called the speech reception threshold (SRT50).
Digits in Noise test (DIN) | Change measures: 0 months, 12 months, 24 months
  A Speech-in-Noise test, validated for the Finnish language. The word material of the test consists of digit triplets presented under stationary background noise (65dB SPL). The result of the DIN is the signal-to-noise ratio at which the participant identifies 50% of the presented triplets correctly, this is called the speech reception threshold (SRT50).

SECONDARY OUTCOMES:
Speech, Spatial and Quality questionnaires - SSQ | Change measures: 0 months, 12 months, 24 months
  The SSQ questionnaire is a self-reporting hearing questionnaire that comprises 49 questions divided into three subdomains: Speech Perception (SP), Spatial Hearing (SH) and other qualities of Hearing (SQ) (18). The answers are provided on an 11-point Likert scale, ranging from 0 to 10.
Hearing aid usage (self-report and HAs log data) | Change measures: 0 months, 12 months, 24 months
  Usage rates of HAs (hours per day) are regularly checked via the HAs' log-data source and recorded during every clinical visit. In addition, participants' own estimation of usage rates is inquired and recorded.
Listening effort questionnaire | Change measures: 0 months, 12 months, 24 months
  Listening effort will be self-reported by the participant for listening tasks of varying difficulties (i.e., different signal-to-noise ratios) on a 10-point VAS scale.
Response time (DIN test) | Change measures: 0 months, 12 months, 24 months
  Response time for the answers given by the participant will be calculated and recorded automatically
Tinnitus Handicap Inventory (THI) | Change measures: 0 months, 12 months, 24 months
  The THI is a 25-item self-report questionnaire for tinnitus that has Functional, Emotional and Catastrophic subscales. It has excellent convergent validity, construct validity and test-retest reliability. The THI takes 10min to complete. Scoring takes 5 min with a score of 4 for a 'yes', 2 for 'sometimes' and 0 for 'no'.
CERAD-nb (global and domain scores) | Change measures: 0 months, 12 months, 24 months
  The Finnish version of the CERAD (Consortium to Establish a Registry for Alzheimer´s Disease) test battery is recommended for assessment of memory disorders in the national Current Care Guidelines developed by the Finnish Medical Society Duodecim (www.kaypahoito.fi).
Clinical Dementia Rating Sum of Boxes (CDR-SoB) | Change measures: 0 months, 12 months, 24 months
  CDR (Clinical Dementia Rating) is used to assess the influence of cognitive impairment on the ability to conduct everyday activities in people with AD and gives a global clinical impression of the functioning level of the study participant. The assessor will interview the participant regarding their cognitive performance on six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on level of impairment: 0 (none), 0.5 (questionable), 1 (mild dementia), 2 (moderate dementia) or 3 (severe dementia). The total Sum of Boxes ranges from 0 (no impairment) to 18 (severe impairment on all domains).
15D questionnaire | Change measures: 0 months, 12 months, 24 months
  A generic, comprehensive, standardized, self-administered questionnaire of health-related quality of life developed in Finland. It includes 15 questions providing a numerical score for patient-perceived health status. It can be used both as a profile and single index score measure. It is commonly used in Finland to assess quality of life in standard care.
EQ5-D-5L questionnaire | Change measures: 0 months, 12 months, 24 months
  A concise, generic measure of self-reported health which is accompanied by weights reflecting the relative importance to people of different types of health problems
Beck Depression Inventory (BDI) | Change measures: 0 months, 12 months, 24 months
  A short, self-administered questionnaire to quantify psychological and physical symptoms of depression. It includes 21 items, and participants are asked to rate each item using a 4-point Likert scale. The BDI is one of the most frequently used questionnaires for the assessment of depression in clinical practice, including in older adults.
Hearing in real-life environment - HERE | Change measures: 0 months, 12 months, 24 months
  The HERE questionnaire is self-reporting hearing questionnaire validated in Finnish language (28). It includes 15 items with a numeric rating scale from 0 to 10 for each item and allows the assessment of hearing with and without hearing aids.

OTHER OUTCOMES:
EEG-derived cortical auditory evoked potentials (CAEPs) | Change measures: 0 months, 12 months, 24 months
  The possible cortical changes related to the use of HA will be measured through EEG-derived cortical auditory evoked potentials (CAEPs) assessed while administering the DIN test.
Structural MRI | Change measures: 0 months, 12 months, 24 months
  sMRI will provide measures of neurodegeneration (e.g., cortical thickness, brain volumes) and cerebrovascular pathology (e.g., white matter lesions, clinically "silent" infarcts). The scans will include T1, T2, FLAIR, and diffusion weighted sequences (~45 min).
Functional MRI | Change measures: 0 months, 12 months, 24 months
  Task-based fMRI scans (~20 min) will be conducted on at least of 30 participants from both groups (60 altogether) closely mimicking the EEG-paradigm (section 3.3.1). To minimize the possible masking effect of scanner noise, the sounds will be presented during silent periods between scans.
Ultra-short echo time MRI / Zero echo time MRI | Change measures: 0 months, 12 months, 24 months
  Task-based ultra-short- and zero echo time MRIs (UTE, ZTE) (~20 min) will also be conducted on the same group of participants having the fMRI described previously. The tasks will closely mimic the EEG-paradigm (section 3.3.1). Short echo time sequences are less sensitive to susceptibility and motion artifacts and the sequences are silent.
Measures related to active lifestyle | Change measures: 0 months, 12 months, 24 months
  Participants will receive a self-administered questionnaire covering several lifestyle domains potentially affected by HI and relevant for dementia risk, e.g. physical, cognitive and social activities. An active lifestyle index will be calculated as a composite score based on these domains.
Digital cognitive test battery | Change measures: 0 months, 12 months, 24 months
  The cognitive test battery includes tests covering different cognitive domains, and available within the public domain. It was adapted and already tested for persons with HI by Prof. Vincent Lin at Sunny Brook University Hospital, Canada, by converting all original verbal instructions into a visual PowerPoint presentation shown on a computer screen. In the HAHA trial, the cognitive test battery will be self-administered by the participant on the DigiKuulo screen at the study site.
1: Vision-related outcomes | Change measures: 0 months, 24 months
  Best-corrected visual acuity
2: Vision-related outcomes | Change measures: 0 months, 24 months
  Slit-lamp examination
3: Vision-related outcomes | Change measures: 0 months, 24 months
  Retinal imaging
4: Vision-related outcomes | Change measures: 0 months, 24 months
  Eye geometrics and biometric values
Blood samples | Change measures: 0 months, 24 months
  Frozen and stored for future assessment of HI or dementia- related markers (e.g. genetic, amyloid, tau, neurodegeneration)
Intervention-related acitivities, intervention group | Change measures: 0 months, 3 months, 6 months, 12 months
  Amplification of HAs
Intervention-related acitivities, standard group | Change measures: 0 months
  Amplification of HAs

CONTACTS AND LOCATIONS:
Overall Officials: Aarno Dietz, prof., Principal Investigator — Kuopio University Hospital and University of Eastern Finland; Alina Solomon, prof., Principal Investigator — University of Eastern Finland
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: Yes
The HAHA Steering Committee and Management Group are open to requests from external researchers for data collected in this study. Applicants will be asked to submit a study protocol, including the research question, planned analysis, and data required. Committee will evaluate this plan (i.e., relevance of the research question, suitability of data, quality of proposed analyses, planned/ongoing HAHA analyses, and other matters) on a case-by-case basis and provide the data or reject the request. Shared data will encompass the data dictionary and de-identified data only. Any analysis will be conducted in collaboration with the HAHA Management Group. Access is subject to the HAHA legal framework. An access agreement will be prepared and signed by both parties.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The trial Steering Committee and Management Group will consider applications for data after the trials results have been published and data will be made available according to the terms of the access agreement.
Access Criteria: As described above in the Plan Description.

REFERENCES:
- [Background] GBD 2019 Hearing Loss Collaborators. Hearing loss prevalence and years lived with disability, 1990-2019: findings from the Global Burden of Disease Study 2019. Lancet. 2021 Mar 13;397(10278):996-1009. doi: 10.1016/S0140-6736(21)00516-X. PMID 33714390
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Brewster KK, Deal JA, Lin FR, Rutherford BR. Considering hearing loss as a modifiable risk factor for dementia. Expert Rev Neurother. 2022 Sep;22(9):805-813. doi: 10.1080/14737175.2022.2128769. Epub 2022 Sep 27. PMID 36150235
- [Background] Sanders ME, Kant E, Smit AL, Stegeman I. The effect of hearing aids on cognitive function: A systematic review. PLoS One. 2021 Dec 31;16(12):e0261207. doi: 10.1371/journal.pone.0261207. eCollection 2021. PMID 34972121
- [Background] Lin MY, Gutierrez PR, Stone KL, Yaffe K, Ensrud KE, Fink HA, Sarkisian CA, Coleman AL, Mangione CM; Study of Osteoporotic Fractures Research Group. Vision impairment and combined vision and hearing impairment predict cognitive and functional decline in older women. J Am Geriatr Soc. 2004 Dec;52(12):1996-2002. doi: 10.1111/j.1532-5415.2004.52554.x. PMID 15571533
- [Background] Gadkaree SK, Sun DQ, Li C, Lin FR, Ferrucci L, Simonsick EM, Agrawal Y. Does Sensory Function Decline Independently or Concomitantly with Age? Data from the Baltimore Longitudinal Study of Aging. J Aging Res. 2016;2016:1865038. doi: 10.1155/2016/1865038. Epub 2016 Sep 27. PMID 27774319
- [Background] Hong T, Mitchell P, Burlutsky G, Liew G, Wang JJ. Visual Impairment, Hearing Loss and Cognitive Function in an Older Population: Longitudinal Findings from the Blue Mountains Eye Study. PLoS One. 2016 Jan 25;11(1):e0147646. doi: 10.1371/journal.pone.0147646. eCollection 2016. PMID 26808979
- [Background] Brenowitz WD, Kaup AR, Lin FR, Yaffe K. Multiple Sensory Impairment Is Associated With Increased Risk of Dementia Among Black and White Older Adults. J Gerontol A Biol Sci Med Sci. 2019 May 16;74(6):890-896. doi: 10.1093/gerona/gly264. PMID 30452551
- [Background] Campbell J, Sharma A. Cross-modal re-organization in adults with early stage hearing loss. PLoS One. 2014 Feb 28;9(2):e90594. doi: 10.1371/journal.pone.0090594. eCollection 2014. PMID 24587400
- [Background] Tarawneh HY, Menegola HK, Peou A, Tarawneh H, Jayakody DMP. Central Auditory Functions of Alzheimer's Disease and Its Preclinical Stages: A Systematic Review and Meta-Analysis. Cells. 2022 Mar 16;11(6):1007. doi: 10.3390/cells11061007. PMID 35326458
- [Background] Davis A, Smith P, Ferguson M, Stephens D, Gianopoulos I. Acceptability, benefit and costs of early screening for hearing disability: a study of potential screening tests and models. Health Technol Assess. 2007 Oct;11(42):1-294. doi: 10.3310/hta11420. PMID 17927921
- [Background] Timmer BHB, Hickson L, Launer S. Do Hearing Aids Address Real-World Hearing Difficulties for Adults With Mild Hearing Impairment? Results From a Pilot Study Using Ecological Momentary Assessment. Trends Hear. 2018 Jan-Dec;22:2331216518783608. doi: 10.1177/2331216518783608. PMID 29956590
- [Background] Wright D, Gagne JP. Acclimatization to Hearing Aids by Older Adults. Ear Hear. 2021 Jan/Feb;42(1):193-205. doi: 10.1097/AUD.0000000000000913. PMID 32769437
- [Background] Panza F, Lozupone M, Solfrizzi V, Sardone R, Dibello V, Di Lena L, D'Urso F, Stallone R, Petruzzi M, Giannelli G, Quaranta N, Bellomo A, Greco A, Daniele A, Seripa D, Logroscino G. Different Cognitive Frailty Models and Health- and Cognitive-related Outcomes in Older Age: From Epidemiology to Prevention. J Alzheimers Dis. 2018;62(3):993-1012. doi: 10.3233/JAD-170963. PMID 29562543
- [Background] Yeo BSY, Song HJJMD, Toh EMS, Ng LS, Ho CSH, Ho R, Merchant RA, Tan BKJ, Loh WS. Association of Hearing Aids and Cochlear Implants With Cognitive Decline and Dementia: A Systematic Review and Meta-analysis. JAMA Neurol. 2023 Feb 1;80(2):134-141. doi: 10.1001/jamaneurol.2022.4427. PMID 36469314
- [Background] Lin FR, Pike JR, Albert MS, Arnold M, Burgard S, Chisolm T, Couper D, Deal JA, Goman AM, Glynn NW, Gmelin T, Gravens-Mueller L, Hayden KM, Huang AR, Knopman D, Mitchell CM, Mosley T, Pankow JS, Reed NS, Sanchez V, Schrack JA, Windham BG, Coresh J; ACHIEVE Collaborative Research Group. Hearing intervention versus health education control to reduce cognitive decline in older adults with hearing loss in the USA (ACHIEVE): a multicentre, randomised controlled trial. Lancet. 2023 Sep 2;402(10404):786-797. doi: 10.1016/S0140-6736(23)01406-X. Epub 2023 Jul 18. PMID 37478886
- [Background] Dietz A, Heinrich A, Tormakangas T, Iso-Mustajarvi M, Miettinen P, Willberg T, Linder PH. The Effectiveness of Unilateral Cochlear Implantation on Performance-Based and Patient-Reported Outcome Measures in Finnish Recipients. Front Neurosci. 2022 Jun 6;16:786939. doi: 10.3389/fnins.2022.786939. eCollection 2022. PMID 35733938
- [Background] Karawani H, Jenkins K, Anderson S. Restoration of sensory input may improve cognitive and neural function. Neuropsychologia. 2018 Jun;114:203-213. doi: 10.1016/j.neuropsychologia.2018.04.041. Epub 2018 May 2. PMID 29729278
- [Background] Glick H, Sharma A. Cross-modal plasticity in developmental and age-related hearing loss: Clinical implications. Hear Res. 2017 Jan;343:191-201. doi: 10.1016/j.heares.2016.08.012. Epub 2016 Sep 6. PMID 27613397
- [Background] Gommeren H, Bosmans J, Cardon E, Mertens G, Cras P, Engelborghs S, Van Ombergen A, Gilles A, Lammers M, Van Rompaey V. Cortical Auditory Evoked Potentials in Cognitive Impairment and Their Relevance to Hearing Loss: A Systematic Review Highlighting the Evidence Gap. Front Neurosci. 2021 Nov 18;15:781322. doi: 10.3389/fnins.2021.781322. eCollection 2021. PMID 34867176
- [Background] Pereira-Jorge MR, Andrade KC, Palhano-Fontes FX, Diniz PRB, Sturzbecher M, Santos AC, Araujo DB. Anatomical and Functional MRI Changes after One Year of Auditory Rehabilitation with Hearing Aids. Neural Plast. 2018 Sep 10;2018:9303674. doi: 10.1155/2018/9303674. eCollection 2018. PMID 30275823
- [Background] Cheung CY, Mok V, Foster PJ, Trucco E, Chen C, Wong TY. Retinal imaging in Alzheimer's disease. J Neurol Neurosurg Psychiatry. 2021 Sep;92(9):983-994. doi: 10.1136/jnnp-2020-325347. Epub 2021 Jun 9. PMID 34108266
- [Background] Solomon A, Stephen R, Altomare D, Carrera E, Frisoni GB, Kulmala J, Molinuevo JL, Nilsson P, Ngandu T, Ribaldi F, Vellas B, Scheltens P, Kivipelto M; European Task Force for Brain Health Services. Multidomain interventions: state-of-the-art and future directions for protocols to implement precision dementia risk reduction. A user manual for Brain Health Services-part 4 of 6. Alzheimers Res Ther. 2021 Oct 11;13(1):171. doi: 10.1186/s13195-021-00875-8. PMID 34635167
- [Background] Dietz A, Buschermohle M, Aarnisalo AA, Vanhanen A, Hyyrynen T, Aaltonen O, Lopponen H, Zokoll MA, Kollmeier B. The development and evaluation of the Finnish Matrix Sentence Test for speech intelligibility assessment. Acta Otolaryngol. 2014 Jul;134(7):728-37. doi: 10.3109/00016489.2014.898185. Epub 2014 May 7. PMID 24807850
- [Background] Smits C, Kapteyn TS, Houtgast T. Development and validation of an automatic speech-in-noise screening test by telephone. Int J Audiol. 2004 Jan;43(1):15-28. doi: 10.1080/14992020400050004. PMID 14974624
- [Background] Willberg T, Buschermohle M, Sivonen V, Aarnisalo AA, Lopponen H, Kollmeier B, Dietz A. The development and evaluation of the Finnish digit triplet test. Acta Otolaryngol. 2016 Oct;136(10):1035-40. doi: 10.1080/00016489.2016.1175662. Epub 2016 Apr 28. PMID 27121373
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Berg L. Clinical Dementia Rating (CDR). Psychopharmacol Bull. 1988;24(4):637-9. No abstract available. PMID 3249765
- [Background] Sintonen H. The 15D instrument of health-related quality of life: properties and applications. Ann Med. 2001 Jul;33(5):328-36. doi: 10.3109/07853890109002086. PMID 11491191
- [Background] Renvall H, Seol J, Tuominen R, Sorger B, Riecke L, Salmelin R. Selective auditory attention within naturalistic scenes modulates reactivity to speech sounds. Eur J Neurosci. 2021 Nov;54(10):7626-7641. doi: 10.1111/ejn.15504. Epub 2021 Nov 3. PMID 34697833
- [Background] Renvall H, Formisano E, Parviainen T, Bonte M, Vihla M, Salmelin R. Parametric merging of MEG and fMRI reveals spatiotemporal differences in cortical processing of spoken words and environmental sounds in background noise. Cereb Cortex. 2012 Jan;22(1):132-43. doi: 10.1093/cercor/bhr095. Epub 2011 May 25. PMID 21613467
- See also: WORLD REPORT ON HEARING — https://youtu.be/EmXwAnP9puQ
- See also: Development of the "Hearing In Real-Life Environments" Questionnaire — http://links.lww.com/EANDH/
- See also: Methods for Analysing and Reporting EQ-5D Data [Internet]. Cham (CH): Springer; 2020. Chapter 1, An Introduction to EQ-5D Instruments and Their Applications — https://www.ncbi.nlm.nih.gov/books/NBK565680/